CLINICAL TRIAL: NCT01821833
Title: A Pilot Randomized, Placebo Controlled, Double Blind Study of Omega-3 Fatty Acids to Prevent Paclitaxel Associated Acute Pain Syndrome
Brief Title: Omega-3 Fatty Acid in Treating Pain in Patients With Breast or Ovarian Cancer Receiving Paclitaxel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New Mexico Cancer Research Alliance (Other)
Collaborators: Alliance Healthcare Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: INST 1211; NCI-2013-00443 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2013-03-27; First posted 2013-04-01 (Estimated); Last update posted 2022-10-05 (Actual); Status verified 2022-10

CONDITIONS: Breast Cancer; Ovarian Neoplasm; Pain
Keywords: omega-3; fatty acids; paclitaxel; acute pain syndrome; peripheral neuropathy; chemotherapy induced neuropathy
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms; Pain; Peripheral Nervous System Diseases | interventions — Fatty Acids, Omega-3; Fish Oils; Omacor; Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Omega-3 fatty acid) (Experimental): Four Omega-3 fatty acid capsules (at 1 gram/capsule) are administered orally daily.
  The capsules may be administered either once daily or as 2 capsules two times daily.
  Interventions: Dietary Supplement: Omega-3 fatty acid; Drug: Paclitaxel
- Arm II (placebo) (Placebo Comparator): Four placebo capsules (at 1 gram microcrystalline cellulose/capsule) are administered orally daily.
  The capsules may be administered either once daily or as 2 capsules two times daily.
  Interventions: Dietary Supplement: Placebo; Drug: Paclitaxel

INTERVENTIONS:
Dietary Supplement: Omega-3 fatty acid — Patients receive omega-3 fatty acid capsules orally beginning 1 week prior to paclitaxel treatment.
  Capsule administration continues until paclitaxel is discontinued or for 12 weeks maximum (whichever comes first).
  Each 1-gram capsule contains approximately 465 mg eicosapentaenoic acid (EPA) and 375 mg docosahexaenoic acid (DHA).
  Other Names: Fish oil; n-3 fatty acid; O3FA; Lovaza
  Arms: Arm I (Omega-3 fatty acid)
Dietary Supplement: Placebo — Patients receive placebo capsules orally beginning 1 week prior to paclitaxel treatment.
  Capsule administration continues until paclitaxel is discontinued or for 12 weeks maximum (whichever comes first)
  Arms: Arm II (placebo)
Drug: Paclitaxel — Patients will receive, as part of their standard of care, weekly paclitaxel at 70 to 90 mg/m2 intravenously for a minimum of 2 months. Treatment 3 out of 4 weeks is allowed.
  Other Names: Taxol

SUMMARY:
Paclitaxel, a widely used chemotherapeutic agent, is associated with several well-known side effects including neuropathy (weakness, numbness and pain) and generalized body aches. The latter has recently been described as paclitaxel-associated acute pain syndrome (P-APS) and often occurs in the first three to four days after administration. It affects about 58-90% of patients. Currently, the mechanism of P-APS is unknown, and there is no standard of care to treat it. However, an intervention with both anti-inflammatory as well as neuroprotective properties would be an ideal candidate for testing in the prevention of P-APS and subsequent development of peripheral neuropathy. Previous studies have suggested that omega-3 fatty acids may act as neuroprotective agents, and there are no currently documented safety concerns with their combined use with paclitaxel.

Therefore, this randomized pilot clinical trial will determine whether omega-3 fatty acids can treat pain in patients with breast or ovarian cancer receiving paclitaxel.

DETAILED DESCRIPTION:
One mechanism proposed for P-APS is an early inflammatory process characterized by macrophage activation in both the dorsal root ganglia and peripheral nerve occurring shortly after paclitaxel therapy. Morphologic alterations in DRG satellite cells have been noted and upregulation of proinflammatory cytokines have been hypothesized as early events in the development of neuropathy. Therefore, it is possible that paclitaxel-induced neuropathic pain may be mediated by pro-inflammatory cytokines. If P-APS and chronic neuropathy are indeed part of a continuum, the inflammatory pathway would be a reasonable target for therapy. While the mechanism of how paclitaxel leads to the development of neuropathy is still not understood, it has been hypothesized that its microtubule-stabilizing effects disrupt axonal transport. Intervention with an agent that is both anti-inflammatory as well as neuroprotective is therefore worth exploring.

Long chain omega-3 fatty acids eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA), are common dietary supplements. They have well established anti-inflammatory properties which serve as the basis for their use in therapeutic trials in inflammatory conditions. Omega -3 fatty acids consumption can attenuate the production of pro-inflammatory metabolites. In addition, it can generate local mediators that facilitate resolution of inflammation. Thus, if P-APS is indeed mediated by inflammation, the anti-inflammatory activity of omega 3 fatty acids may be one mechanism to prevent P-APS. Additionally, given its well established safety profile, it may be an attractive alternative to NSAIDS.

A dose of at least 2.7 g/day of EPA and DHA have been reported to have analgesic effects in inflammatory conditions. The dose of 4 g/day is an FDA-approved dose of omega 3 fatty acids (Lovaza) for the treatment of hypertriglyceridemia and has a well-documented toxicity profile. On the basis of this, a dose of 4 g/day was selected for this study. Lovaza (omega-3-acid ethyl esters) capsules will be used. Each 1-gram capsule contains approximately 465 mg EPA and 375 mg DHA.

ELIGIBILITY:
Inclusion Criteria:

* Patients have a diagnosis of breast cancer or ovarian cancer
* Patients are scheduled to receive weekly paclitaxel at 70-90 mg/m^2 for a minimum of 2 months; 3 out of 4 weeks is allowed
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0, 1 or 2
* Patients must not have taken omega-3-fatty acid supplements within the past 1 month prior to registration and must agree to refrain from use of omega- 3 fatty acid supplements from sources outside the study
* Patients must not be on nonsteroidal anti-inflammatory drugs (NSAIDS) or aspirin for at least 1 week prior to registration; NSAIDS or aspirin are allowed after enrollment
* Patients must not have received any other analgesics (opiates and tramadol) 1 week prior to registration; analgesics (opiates and tramadol) are allowed after enrollment
* Patients must have the ability to complete questionnaires by themselves or with assistance
* Patients must not be on anticoagulation medication (heparin/ warfarin) within 28 days prior to registration, because of increased risk of bleeding
* Concurrent treatment with carboplatin +/- bevacizumab is allowed
* Concurrent treatment with human epidermal growth factor receptor (Her2 neu) targeted therapy is allowed

Exclusion Criteria:

* Known allergy to omega 3 fatty acids, fish or shellfish
* Pre-existing diagnosis of peripheral neuropathy
* Diagnosis of fibromyalgia
* Concurrent planned neutrophil colony stimulating factor therapy
* Prior exposure to paclitaxel within the last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-05-24 (Actual); Primary Completion 2018-01-16 (Actual); Study Completion 2022-08-03 (Actual)

PRIMARY OUTCOMES:
Mean severity of pain | Up to 1 month after completion of therapy
  Differences between groups will analyzed via t-tests or Wilcoxon rank-sum tests as appropriate.

SECONDARY OUTCOMES:
Incidence of pain or relief | Up to 1 month after completion of therapy
  Fisher's exact test will be used for the incidence variable with 95% confidence intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Zoneddy Dayao, Principal Investigator — University of New Mexico Comprehensive Cancer Center
Locations (2):
- United States (2):
  - University of New Mexico Comprehensive Cancer Center, Albuquerque, New Mexico
  - Presbyterian Medical Group, Albuquerque, New Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tawfik B, Dayao ZR, Brown-Glaberman UA, Pankratz VS, Lafky JM, Loprinzi CL, Barton DL. A pilot randomized, placebo-controlled, double-blind study of omega-3 fatty acids to prevent paclitaxel-associated acute pain syndrome in breast cancer patients: Alliance A22_Pilot2. Support Care Cancer. 2023 Oct 17;31(12):637. doi: 10.1007/s00520-023-08082-x. PMID 37847317
- See also: University of New Mexico Cancer Center — http://cancer.unm.edu
- See also: New Mexico Cancer Care Alliance — http://www.nmcca.org

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-01): https://cdn.clinicaltrials.gov/large-docs/33/NCT01821833/Prot_SAP_000.pdf